CLINICAL TRIAL: NCT03311412
Title: A Phase 1, Open-Label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Antineoplastic Activity of Sym021 (Anti-PD-1) as Monotherapy, in Combination With Either Sym022 (Anti-LAG-3) or Sym023 (Anti-TIM-3), and in Combination With Both Sym022 and Sym023 in Patients With Advanced Solid Tumor Malignancies or Lymphomas
Brief Title: Sym021 Monotherapy, in Combination With Sym022 or Sym023, and in Combination With Both Sym022 and Sym023 in Patients With Advanced Solid Tumor Malignancies or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Sym021-01
Record Dates: First submitted 2017-10-03; First posted 2017-10-17 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Cancer; Solid Tumor; Lymphoma
Keywords: Locally advanced/unresectable; Metastatic solid tumor; Lymphoma; Anti-PD-1; PD-1; PD1; Anti-LAG-3; LAG-3; LAG3; Anti-TIM-3; TIM-3; TIM3
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Sym021 Dose Level 1 (Experimental): Part 1, Sym021 monotherapy dose level 1
  Interventions: Drug: Sym021
- Sym021 Dose Level 2 (Experimental): Part 1, Sym021 monotherapy dose level 2
  Interventions: Drug: Sym021
- Sym021 Dose Level 3 (Experimental): Part 1, Sym021 monotherapy dose level 3
  Interventions: Drug: Sym021
- Arm A: Sym021+Sym022 Dose Level 1 (Experimental): Part 2, Arm A: Sym021 RP2D in combination with dose level 1 of Sym022
  Interventions: Drug: Sym021; Drug: Sym022
- Arm A: Sym021+Sym022 Dose Level 2 (Experimental): Part 2, Arm A: Sym021 RP2D in combination with dose level 2 of Sym022
  Interventions: Drug: Sym021; Drug: Sym022
- Arm A: Sym021+Sym022 Dose Level 3 (Experimental): Part 2, Arm A: Sym021 RP2D in combination with dose level 3 of Sym022
  Interventions: Drug: Sym021; Drug: Sym022
- Arm A: Sym021+Sym022 Dose Level 4 (Experimental): Part 2, Arm A: Sym021 RP2D in combination with dose level 4 of Sym022
  Interventions: Drug: Sym021; Drug: Sym022
- Arm B: Sym021+Sym023 Dose Level 1 (Experimental): Part 2, Arm B: Sym021 RP2D in combination with dose level 1 of Sym023
  Interventions: Drug: Sym021; Drug: Sym023
- Arm B: Sym021+Sym023 Dose Level 2 (Experimental): Part 2, Arm B: Sym021 RP2D in combination with dose level 2 of Sym023
  Interventions: Drug: Sym021; Drug: Sym023
- Arm B: Sym021+Sym023 Dose Level 3 (Experimental): Part 2, Arm B: Sym021 RP2D in combination with dose level 3 of Sym023
  Interventions: Drug: Sym021; Drug: Sym023
- Arm B: Sym021+Sym023 Dose Level 4 (Experimental): Part 2, Arm B: Sym021 RP2D in combination with dose level 4 of Sym023
  Interventions: Drug: Sym021; Drug: Sym023
- Arm B: Sym021+Sym023 Dose Level 5 (Experimental): Part 2, Arm B: Sym021 RP2D in combination with dose level 5 of Sym023
  Interventions: Drug: Sym021; Drug: Sym023
- Sym021+Sym022+Sym023 Dose Level 1 (Experimental): Part 3, Sym021 in combination with Sym022 and Sym023
  Interventions: Drug: Sym021; Drug: Sym022; Drug: Sym023
- Sym021+Sym022+Sym023 Dose Level 2 (Experimental): Part 3, Sym021 in combination with Sym022 and Sym023
  Interventions: Drug: Sym021; Drug: Sym022; Drug: Sym023
- Sym021+Sym022+Sym023 Dose Level 3 (Experimental): Part 3, Sym021 in combination with Sym022 and Sym023
  Interventions: Drug: Sym021; Drug: Sym022; Drug: Sym023
- Sym021+Sym022+Sym023 Dose Level 4 (Experimental): Part 3, Sym021 in combination with Sym022 and Sym023
  Interventions: Drug: Sym021; Drug: Sym022; Drug: Sym023
- Sym021+Sym022+Sym023 Dose Level 5 (Experimental): Part 3, Sym021 in combination with Sym022 and Sym023
  Interventions: Drug: Sym021; Drug: Sym022; Drug: Sym023

INTERVENTIONS:
Drug: Sym021 — Sym021 is a humanized antibody that binds PD-1 with sub-nanomolar affinity and blocks binding of the inhibitory ligands PD-L1 and PD-L2, thus releasing PD-1-mediated inhibition of the immune response.
  Other Names: Anti-PD-1
Drug: Sym022 — Sym022 is a recombinant, fully human antibody that binds LAG-3 and blocks the LAG-3/major histocompatibility complex class II (MHC-II) interaction, thus allowing for increased T-cell proliferation and cytokine production.
  Other Names: Anti-LAG-3
  Arms: Arm A: Sym021+Sym022 Dose Level 1; Arm A: Sym021+Sym022 Dose Level 2; Arm A: Sym021+Sym022 Dose Level 3; Arm A: Sym021+Sym022 Dose Level 4; Sym021+Sym022+Sym023 Dose Level 1; Sym021+Sym022+Sym023 Dose Level 2; Sym021+Sym022+Sym023 Dose Level 3; Sym021+Sym022+Sym023 Dose Level 4; Sym021+Sym022+Sym023 Dose Level 5
Drug: Sym023 — Sym023 is a recombinant, fully human antibody that binds TIM-3 and induces activation of immune cells.
  Other Names: Anti-TIM-3
  Arms: Arm B: Sym021+Sym023 Dose Level 1; Arm B: Sym021+Sym023 Dose Level 2; Arm B: Sym021+Sym023 Dose Level 3; Arm B: Sym021+Sym023 Dose Level 4; Arm B: Sym021+Sym023 Dose Level 5; Sym021+Sym022+Sym023 Dose Level 1; Sym021+Sym022+Sym023 Dose Level 2; Sym021+Sym022+Sym023 Dose Level 3; Sym021+Sym022+Sym023 Dose Level 4; Sym021+Sym022+Sym023 Dose Level 5

SUMMARY:
The primary purpose of this study is to see if Sym021 is safe and tolerable as monotherapy, in combination with either Sym022 or Sym023, and in Combination with both Sym022 and Sym023 for patients with locally advanced/unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available.

DETAILED DESCRIPTION:
Part 1 of this study will evaluate the safety, tolerability, and dose-limiting toxicities (DLTs) to establish the maximum tolerated dose (MTD) and/or the selected dose of sequential escalating doses of Sym021 when administered once every 2 weeks (Q2W) by IV infusion to patient cohorts with locally advanced/unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available

Part 2 of the study will evaluate the safety, tolerability, and DLTs to establish the MTD and/or the selected dose of sequential escalating doses of Sym022 when administered Q2W in combination with a fixed dose of 3 mg/kg of Sym021, each by IV infusion to patient cohorts with locally advanced/unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available

Part 3 of the study will evaluate of the safety, tolerability, and DLTs to establish the MTD and/or the selected dose of sequential escalating doses of Sym023 when administered Q2W in combination with fixed doses of 3 mg/kg of Sym021 and either 1, 3 or 5 mg/kg of Sym022, each by IV infusion to patient cohorts with locally advanced/unresectable or metastatic solid tumor malignancies or lymphomas that are refractory to available therapy or for which no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age at the time of obtaining informed consent.
* Documented (histologically- or cytologically-proven) solid tumor malignancy that is locally advanced or metastatic; patients with documented lymphoma.
* Malignancy (solid tumor or lymphoma) that is currently not amenable to surgical intervention due to either medical contraindications or non-resectability of the tumor.
* Refractory to or intolerant of existing therapy(ies) known to provide clinical benefit.
* Measurable or non-measurable disease according to RECIST v1.1 or RECIL 2017.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Persons of childbearing potential agreeing to use a highly effective method of contraception during the study beginning within 2 weeks prior to the first dose and continuing until 6 months after the last dose of study drug(s); men agreeing to refrain from sperm donation during this period.

Exclusion Criteria:

* Women who are pregnant or intending to become pregnant before, during, or within 6 months after the last dose of study drug; women who are breastfeeding; persons of childbearing potential and not willing to use a highly effective method of contraception.
* Central nervous system (CNS) malignancies; patients with known, untreated CNS or leptomeningeal metastases, or spinal cord compression, patients with any of the above not controlled by prior surgery or radiotherapy, or patients with symptoms suggesting CNS involvement for which treatment is required.
* Hematologic malignancies other than lymphoma.
* Active thrombosis, or a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within 4 weeks prior to Cycle 1/Day 1 (C1/D1) unless adequately treated and considered stable.
* Active uncontrolled bleeding or a known bleeding diathesis.
* Clinically significant cardiovascular disease or condition.
* Significant ocular disease or condition, including history of an autoimmune or inflammatory disorder.
* Significant pulmonary disease or condition.
* Current or recent (within 6 months) significant gastrointestinal (GI) disease or condition.
* An active, known, or suspected autoimmune disease, or a documented history of autoimmune disease or syndrome, requiring systemic steroids or other immunosuppressive medications.
* History of organ transplantation (e.g., stem cell or solid organ transplant).
* History of significant toxicities associated with previous administration of immune checkpoint inhibitors that necessitated permanent discontinuation of that therapy.
* Patients with unresolved > Grade 1 toxicity associated with any prior antineoplastic therapy except for persistent Grade 2 alopecia, peripheral neuropathy, decreased hemoglobin, lymphopenia, hypomagnesemia, and/or end-organ failure being adequately managed by hormone replacement therapy.
* Inadequate recovery from any prior surgical procedure, or having undergone any major surgical procedure within 4 weeks prior to C1/D1.
* Known history of human immunodeficiency virus (HIV) or known active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).

Drugs and Other Treatments Exclusion Criteria:

* Part 2 Combination Dose-Escalations ONLY: Prior therapy with:

  * Sym021 or other inhibitors of PD-1/PD-L1.
  * Sym022 or other inhibitors of LAG-3, if participating in Arm A.
  * Sym023 or other inhibitors of TIM-3, if participating in Arm B.
* Part 3 Combination Dose-Escalations ONLY: Prior therapy with:

  * Sym022 or other inhibitors of LAG-3
  * Sym023 or other inhibitors of TIM-3
* Any antineoplastic agent for the primary malignancy (standard or investigational) within 4 weeks or 5 plasma half-lives, whichever is shortest, prior to first study drug administration and during study, with exceptions.
* Any other investigational treatments within 2 weeks prior to and during study; includes participation in any medical device or supportive care therapeutic intervention trials.
* Radiotherapy, with exceptions.
* Use of live vaccines against infectious diseases 4 weeks prior to first study drug administration and during study.
* Immunosuppressive or systemic hormonal therapy within 2 weeks prior to first study drug administration and during study, with exceptions.
* Prophylactic use of hematopoietic growth factors within 1 week prior to first study drug administration and during Cycle 1 of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Part 1: Assessment of treatment emergent adverse events (AEs) meeting DLT criteria. | 12 months
  Assess the safety and tolerability of Sym021 monotherapy on a Q2W schedule. Assessment based on the occurrence of AEs meeting DLT criteria measured during Cycle 1.
Part 2: Assessment of treatment emergent adverse events (AEs) meeting DLT criteria. | 12 months
  Assess the safety and tolerability of the Sym021 RP2D in combination with sequential escalating doses of Sym022 or Sym023 on a Q2W schedule. Assessment based on the occurrence of AEs meeting DLT criteria measured during Cycle 1.
Part 3: Assessment of treatment emergent adverse events (AEs) meeting DLT criteria. | 12 months
  Assess the safety and tolerability of the Sym021 RP2D in combination with sequential escalating doses of Sym022 and Sym023 on a Q2W schedule. Assessment based on the occurrence of AEs meeting DLT criteria measured during Cycle 1.

SECONDARY OUTCOMES:
Evaluation of the immunogenicity of Sym021 as a single agent and in combination with Sym022 and Sym023. | 24 months
  Serum sampling to assess the potential for anti-drug antibody (ADA) formation.
Evaluation of objective response (OR) or stable disease (SD). | 24 months
  Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), Response Evaluation Criteria in Lymphomas 2017 (RECIL 2017), or Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST), depending on tumor type.
Time to progression (TTP) of disease. | 24 months
  Based on time of enrollment to first evidence of progression on imaging studies, as assessed by RECIST v1.1, RECIL 2017, or iRECIST, depending on tumor type.
Area under the concentration-time curve in a dosing interval (AUC) | 24 months
  Will be estimated using non-compartmental methods and actual timepoints.
Maximum concentration (Cmax) | 24 months
  Will be derived from observed data.
Time to reach maximum concentration (Tmax) | 24 months
  Will be derived from observed data.
Trough concentration (Ctrough) | 24 months
  Will be derived from observed data.
Terminal elimination half-life (T½) | 24 months
  Will be estimated using non-compartmental methods and actual timepoints.
Clearance (CL) | 24 months
  Will be estimated using non-compartmental methods and actual timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, FRCPC, Principal Investigator — Princess Margaret Cancer Centre
Locations (4):
- United States (3):
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No